CLINICAL TRIAL: NCT05931003
Title: Reconstruction of the Carotid Bifurcation in Patients With Arterial Hypertension of 2-3 Degrees
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samara State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hypertension_after_CEA_or_CAS
Record Dates: First submitted 2023-04-15; First posted 2023-07-05 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hypertension; Carotid Stenosis; Symptomatic Carotid Artery Stenosis
Keywords: Hypertension; Carotid Stenosis; Symptomatic Carotid Artery Stenosis; Glomus ectomy; Carotid endarterectomy; Carotid Stenting
MeSH Terms: conditions — Hypertension; Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carotid artery stenting (Experimental): Carotid artery stenting
  Interventions: Procedure: Carotid stenting
- Carotid endarterectomy (Active Comparator): Carotid endarterectomy
  Interventions: Procedure: Carotid endarterectomy

INTERVENTIONS:
Procedure: Carotid stenting — In carotid stenting, a long, hollow tube (catheter) is threaded through the arteries to the narrowed carotid artery in the neck. A metal mesh tube (stent) is inserted into the vessel to serve as a scaffold that helps prevent the artery from narrowing again. The catheter and the filter - which catches any debris that may break off during the procedure - are removed.
  Arms: Carotid artery stenting
Procedure: Carotid endarterectomy — Carotid endarterectomy is a procedure to treat carotid artery disease. In carotid endarterectomy receive general anesthesia. Surgeon makes an incision along the front of your neck, opens your carotid artery and removes the plaques that are clogging artery. Then, surgeon repairs the artery with stitches or a patch made with a vein or artificial material (patch graft).
  Sometimes surgeons may use another technique called eversion carotid endarterectomy. This involves cutting the carotid artery and turning it inside out, then removing the plaque. Surgeon then reattaches the artery.
  Arms: Carotid endarterectomy

SUMMARY:
Carotid endarterectomy (CEA) is a well-established procedure for preventing ischemic brain damage. Stenosis of the precerebral vessels are often combined with arterial hypertension. In recent decades, many works have appeared that indicate that the course of arterial hypertension (AH) changes after CEA. However, it remains unknown how this is related to the choice of surgical tactics.

DETAILED DESCRIPTION:
Purpose of the study: to substantiate the choice of the method of surgical treatment in patients with a combination of hemodynamically significant stenosis of the carotid bifurcation and arterial hypertension of 2-3 degrees.

Tasks:

1. To study the course of hypertension after carotid endarterectomy with removal of the carotid glomus.
2. To study the course of hypertension in patients after stenting of the internal carotid artery.
3. To substantiate the strategy for performing carotid endarterectomy in patients with bilateral significant lesions of the internal carotid artery.
4. To substantiate the choice of a surgical treatment strategy in patients with significant stenosis of the carotid bifurcation and 2-3 degree of hypertension.

Methods for examining patients: collection of complaints and anamnesis, objective examination, questioning of patients, instrumental examination (ultrasound of BCS, daily monitoring of blood pressure, CT of the brain, cerebral angiography).

As a result of the study, the optimal tactics of surgical treatment in patients with carotid artery stenosis and the presence of hypertension will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptomatic ICA stenosis 70-90%
* Arterial hypertension of 2 or 3 degrees
* CEA operation with carotid glomus removal or ICA stenting operation

Exclusion Criteria:

* severe diabetes
* traumatic brain injury in history
* IHD, stable angina pectoris 3-4 FC.
* presence of clinical signs of vertebrobasilar insufficiency
* the presence of significant stenosis of the renal arteries
* CKD stages 3b-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change the degree of arterial hypertension | 2 years
  Using ambulatory blood pressure monitoring (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Samara State Medical University, Samara, Russia

REFERENCES:
- See also: ARTERIAL HYPERTENSION AFTER CAROTID ENDARTERECTOMY AND INTERNAL CAROTID ARTERY STENTING — https://www.angiolsurgery.org/magazine/2022/3/